CLINICAL TRIAL: NCT04184583
Title: Registry Study on Drug Therapy and Clinical Outcomes in Patients With Acute Coronary Syndrome
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Lin Yang, Director of pharmacy department of Beijing Anzhen Hospital, Beijing Anzhen Hospital
Other Study IDs: ANZHEN HOSPITOL-LY-02
Record Dates: First submitted 2019-11-28; First posted 2019-12-03 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Drug Therapy; Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Biospecimen Retention: Samples With DNA — Part of DNA samples were preserved in the -80℃.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Registry Study on Drug Therapy and Clinical Outcomes in Patients With Acute Coronary Syndrome

ELIGIBILITY:
Inclusion Criteria:

* Informed consent has been signed.
* Patients diagnosed in our hospital with acute coronary syndrome.
* Age ≥18.
* Life expectancy ≥12 months.

Exclusion Criteria:

* Severe lack of important information such as history of previous medication, history of previous disease, history of surgery.
* Pregnant and lactating women.
* Mental disorders, or inability to communicate effectively with researchers, or failure to comply with research protocols.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Acute Coronary Syndrome with blood concentration monitoring or genetic testing at the pharmacy department of Beijing Anzhen Hospital from January 1, 2018.Those who fill the inclusion criteria at screening will be invited for the registry study into different groups.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
main adverse cardiovascular and cerebrovascular events (MACCE) | up to 5 years
  MACCE will be defined as all-cause death, non-fatal stroke, non-fatal myocardial infarction (MI), and ischemic-driven revascularization.

SECONDARY OUTCOMES:
Adverse drug reaction | up to 5 years
  Adverse drug reaction will be defined as any adverse reactions in the patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital, Beijing, Beijing Municipality, China